CLINICAL TRIAL: NCT07295951
Title: An Open-Label Study to Investigate the Absorption, Metabolism, And Excretion (AME) Of 14C-Bleximenib (JNJ-75276617) in Participants With Acute Leukemia
Brief Title: A Study of 14C-Bleximenib (Radiolabeled) in Participants With Acute Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 75276617ALE1006; 75276617ALE1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Leukemias; Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bleximenib (Experimental): Participants will receive a single oral dose of 14C-bleximenib on Cycle 1 Day 1. The recommended Phase 2 dose (RP2D) of bleximenib will start on Cycle 1 Day 2 with non-radiolabeled bleximenib and will continue until the end of Cycle 1 (cycle duration=28 days), with subsequent roll-over for eligible participants to 75276617ALE1001 (NCT04811560) for continued non-radiolabeled bleximenib administration as appropriate.
  Interventions: Drug: 14C-bleximenib; Drug: bleximenib

INTERVENTIONS:
Drug: 14C-bleximenib — 14C-bleximenib will be administered orally.
  Other Names: JNJ-75276617
Drug: bleximenib — Non-radiolabeled bleximenib will be administered orally.
  Other Names: JNJ-75276617

SUMMARY:
The purpose of this study is to assess how the body absorbs, breaks down (metabolism), and removes (excretes) radiolabeled bleximenib (a drug molecule that has been chemically bonded with a radioactive isotope which emits radiation making it easier to track in the body) in participants with acute leukemia (highly aggressive blood cancer typically characterized by large numbers of immature white blood cells in the bone marrow).

ELIGIBILITY:
Inclusion criteria:

* Body weight greater than or equal to (>=) 40 kilograms (kg)
* Relapsed or refractory (R/R) acute leukemia harboring histone-lysine N-methyltransferase 2A (KMT2A), nucleophosmin 1 (NPM1), nucleoporin 98 (NUP98) or nucleoporin 214 (NUP214) gene alterations, and has exhausted, or is ineligible for available therapeutic options
* Eastern cooperative oncology group (ECOG) performance status grade of 0 or 1
* Regular bowel movements (that is [i.e.], average production of at least one stool every 2 days)
* A woman of childbearing potential must have a negative highly sensitive serum beta-human chorionic gonadotropin at screening and within 48 hours prior to the first dose of study treatment

Exclusion criteria:

* Acute promyelocytic leukemia or diagnosis of Down syndrome associated leukemia, according to world health organization (WHO) 2016 criteria
* Active central nervous system (CNS) disease
* Recipient of solid organ transplant
* Any toxicity (except for alopecia, stable peripheral neuropathy, thrombocytopenia, neutropenia, anemia) from previous anticancer therapy that has not resolved to baseline or to Grade 1 or less
* Major surgery (e.g., requiring general anesthesia) within 2 weeks prior to first dose of study treatment or has not recovered from surgery or has major surgery planned during the time the participant is receiving study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-06-14 (Estimated); Study Completion 2026-07-13 (Estimated)

PRIMARY OUTCOMES:
Percentage of Dose Excreted in Urine (feu) | Up to Day 28
  Total amount excreted into the urine, expressed as a percentage of the administered dose will be reported.
Percentage of Dose Excreted in Feces (fef) | Up to Day 28
  Total amount excreted into the feces expressed as a percentage of the administered dose will be reported.
Amount Excreted in Urine (Aeu) | Up to Day 28
  Aeu defined as the total amount of bleximenib and radioactivity excreted into the urine will be reported.
Amount Excreted in Feces (Aef) | Up to Day 28
  Aef defined as the total amount of bleximenib and radioactivity excreted into the feces will be reported.
Area Under the Concentration-Time Curve from Time 0 to the Last Measurable Concentration (AUC0-t) | Cycle 1 Day 1, and Cycle 1 Day 2 (Cycle duration=28 days)
  AUC0-t in whole blood and plasma will be reported.
Maximum Observed Concentration (Cmax) | Cycle 1 Day 1, and Cycle 1 Day 2 (Cycle duration=28 days)
  Maximum observed concentration in whole blood and plasma will be determined.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 58 days
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the study treatment. A SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- The Christie NHS Foundation Trust Christie Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency